CLINICAL TRIAL: NCT02512432
Title: INTACS (Intrastromal Corneal Ring Segments) For Corneal Ectasia
Acronym: INTACS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Christopher Heichel, MD, Associate Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150826
Record Dates: First submitted 2015-07-29; First posted 2015-07-30 (Estimated); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Keratoconus (Other)
  Interventions: Device: INTACS

INTERVENTIONS:
Device: INTACS — asymmetrical corneal inserts to reduce, or eliminate myopia and astigmatism in patients with keratoconus to decrease dependence on contact lenses and spectacle correction, while potentially deferring need for corneal transplantation.

SUMMARY:
To join established study put on by Addition Technologies, Inc. in the surgical implantation of asymmetrical INTACS segments to treat myopia and astigmatism in patients with keratoconus.

DETAILED DESCRIPTION:
Use of asymmetrical corneal inserts to reduce or eliminate myopia and astigmatism in patients with keratoconus, who are no longer able to achieve adequate vision with their contact lenses or spectacles, so that their functional vision may be restored and the need for corneal transplantation may potentially be deferred.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age, or older
* have experienced a progressive deterioration in their vision, such that they can no longer achieve adequate functional vision on a daily basis with contact lenses, or spectacles.
* have clear central corneas
* have a corneal thickness of 450 microns or greater at the proposed incision site
* have corneal transplantation as the only remaining option to improve their visual function

Exclusion Criteria:

* under 21 years of age
* have not experienced a progressive deterioration in their vision, such that they can no longer achieve adequate functional vision on a daily basis with contact lenses, or spectacles.
* do not have clear central corneas
* do not have a corneal thickness of 450 microns or greater at the proposed incision site
* do not have corneal transplantation as the only remaining option to improve their visual function

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Corneal mapping to measure corneal thickness and steepening | 1 year
  Corneal Topography

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Heichel, MD, Principal Investigator — University of California, San Diego, Shiley Eye Institute